CLINICAL TRIAL: NCT01168882
Title: Phase 1 Open-label, Dose-escalation Clinical Study of the Safety and Tolerability of RGB-286638, a Novel, Multi-targeted Kinase Inhibitor, Administered to Patients With Selected, Relapsed or Refractory Hematological Malignancies
Brief Title: Safety and Tolerability of RGB-286638 in Patients With Selected, Relapsed or Refractory Hematological Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to not initiate clinical trial at this time
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGB638-1-08-02
Record Dates: First submitted 2010-07-20; First posted 2010-07-23 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Hematological Malignancies
Keywords: RGB-286638; Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — RGB 286638

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: RGB-286638 — The starting dose is a flat-fixed dose of 40 mg given i.v. over 60 min, weekly x3, of a 28-days cycle (q4 weeks)

SUMMARY:
The purpose of the study is to determine the safety and tolerability of RGB-286638, a novel, multi-targeted kinase inhibitor, administered to patients with selected, relapsed or refractory hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed diagnosis of:

  * Multiple myeloma (MM)
  * Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL)
  * Mantle Cell Lymphoma (MCL)
  * Chronic Myelogenous Leukemia (CML)
* Refractory to/relapsed after and/or intolerant of one or more standard therapies or for which no standard therapy exists.
* ECOG performance status 0-2.
* Adequate bone marrow, cardiovascular, renal and hepatic function
* Recovery from all adverse events due to prior therapies
* Contraception

Exclusion Criteria:

* Prior chemotherapy, monoclonal antibodies, investigational agents, or radiation therapy (involving ≥ 30% of the active bone marrow) within 14 days prior to the first dose (note nitrosoureas and mitomycin are not permitted for at least 42 days before the first dose of RGB-286638).
* CNS involvement of the hematological malignancy.
* Active or unstable cardiac disease and/or history of myocardial infarction within 6 months and/or history of clinically significant ventricular arrhythmias.
* Concomitant therapies that are known to prolong the QT interval and are associated with a risk of Torsades de Pointes (TdP) are not permitted within 7 days before the first dose; however, amiodarone is not permitted within 90 days before the first dose.
* Patients with uncontrolled and unstable intercurrent illness.
* Concomitant therapy with inhibitors and/or inducers of CYP450 3A4 within 1 week of the first dose.
* Bleeding disorder unrelated to hematological malignant disease.
* HIV or HIV-related malignancy.
* History of other malignancies except: (i) adequately treated basal or squamous cell carcinoma of the skin; (ii) curatively treated, a) in situ carcinoma of the uterine cervix, b) prostate cancer, or c) superficial bladder cancer; or (iii) other curatively treated solid tumor with no evidence of disease for ≥ 2 years.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 Days of Cycle 1

SECONDARY OUTCOMES:
Safety and Tolerability of escalating doses of RGB-286638 | 30 days after the last study drug is given to a subject
  Frequency and Severity of Adverse Events based on NCI Common Terminology Criteria for Adverse Events (CTCAE) v 3.0 (2003)
Objective Tumor Response | At the Time of Final Analysis
Pharmacokinetic Properties | At the end of Cycle 1 (28 days)
Pharmacodynamic properties | At the end of Cycle 1 (28 days)